<u>Study identifiers:</u> DIAD Devic's Disease Auto 2008; NCT00787722 <u>Study title:</u> Hematopoietic Stem Cell Transplant in Devic's Disease

# TRIAL OF HIGH DOSE IMMUNOSUPPRESSIVE THERAPY WITH HEMATOPOIETIC STEM CELL SUPPORT IN DEVIC'S DISEASE

#### Principal Investigator:

Richard K. Burt, M.D., Chief Division of Immunotherapy, Northwestern University, Chicago, USA

# Co-Investigators:

Roumen Balabanov, M.D. Rush University Multiple Scierosis Center, Chicago, USA

Kimberly Yaung Grady, R.N. Division of Immunotherapy, Northwestern University, Chicago, USA

Kate Quigley, R.N., M.B.A. Division of Immunotherapy, Northwestern University, Chicago, USA

Robert Sufit, M.D.

Department of Neurology, Northwestern University, Chicago, USA

#### Statistician:

Borko Jovanovic, Ph.D., Northwestern University, Chicago, USA

# TABLE OF CONTENTS

| 1.0 | Precis | 3 |
|------|-----------------------------------------------------|-----|
| 2.0 | Objectives | 3 |
| 3.0 | Background of Devic's disease | 4 |
| 4.0 | Rationale for the Proposed Treatment and Scientific | |
| | Justification | 7 |
| 5.0 | Eligibility | 10 |
| 6.0 | Treatment Plan | 12 |
| 7.0 | Hospital Discharge Guidelines | 16 |
| 8.0 | Side Effects | 16 |
| | Drug Information | 17 |
| | Evaluation of Toxicity | 18 |
| | Adverse Event Reporting | 19 |
| | Evaluation of Response | 19 |
| | Data Management | 19 |
| | Statistical references | 19 |
| | Criteria for removal from study | 19 |
| | Follow up procedures | 19 |
| 17.0 | | 20 |
| | Records to be kept | 20 |
| | | 21 |
| 20.0 | 11 | 27 |
| | Appendix I: MRC (Medical Research Council) | |
| | Scale | 27 |
| | Appendix II: EDSS (Expanded Disability Status | |
| | Scale) | 28 |
| | Appendix III: NRS (Neurologic Rating Scale) | 34 |
| | Appendix IV: PASAT ( Paced Auditory Serial | |
| | Addition ) | 35 |
| | Appendix V: SF-36 (Social Functioning -36) | 39 |
| | Appendix VI: FACT- BMT (Functional | |
| | Assessment of Cancer Therapy – | 4.0 |
| | Bone Marrow Transplantation ) | 46 |

#### 1.0 Precis

Neuromyelitis optica (NMO, Devic's disease) is an autoimmune, inflammatory, demyelinating central nervous system disorder in which a person's own immune system attacks the optic nerves and spinal cord and is characterized by concurrence of optic neuritis and transverse myelitis, typically associated with a lesion in the spinal cord extending over three or more vertebral segments. Although it is most commonly relapsing, it is distinct from multiple sclerosis in that it is more severe, tends to spare the brain, and is associated with a longitudinally extensive lesion on spinal cord MRI. Furthermore, NMO is associated with a highly specific serum autoantibody marker, NMO-lgG, which targets the water channel aquaporin-4. The disease follows a relapsing course in more than 90% of patients. Vision and ambulation are significantly impaired within 5 years of its onset in approximately half of patients (46). Relapses usually occur early with about 55% of patients having a relapse in the first year and 90% in the first 5 years (47). Unlike MS, Devic's disease rarely has a secondary progressive phase in which patients have increasing neurologic decline between attacks without remission. Instead, disabilities arise from the acute attacks (47).

Approximately 20% of patients with monophasic Devic's disease have permanent visual loss and 30% have permanent paralysis in one or more legs. Among patients with relapsing Devic's disease, 50% have paralysis or blindness within 5 years. In some patients (33% in one study), transverse myelitis in the cervical spinal cord resulted in respiratory failure and subsequent death (47).

At present, parenteral corticosteroids are widely employed as first-line treatment of optic neuritis and myelitis attacks, whereas therapeutic plasmapheresis is applied in the case of corticosteroids failure. Various strategies for the prevention of NMO relapses have been employed in small case series with modest activity. Immune based therapies, in order to be effective, need to be started early in the disease course while Devic's disease is predominantly an immune-mediated and inflammatory disease. Since 50% of patients with NMO are confined to a wheelchair within 5 years of onset, new therapies are needed in this disease.

We now propose, as a phase I study, complete immune ablation and subsequent reconstitution with autologous stem cells.

# 2.0 Objectives

To evaluate the safety (phase I) of autologous hematopoietic stem cell transplantation for inflammatory, autoimmune and demyelinating NMO. The primary endpoints to be considered in this study are:

# 2.1 Primary Endpoint:

- 1. Survival.
- -2. Visual aculty.
- Decreased weakness in limb (MRC) (see appendix).

#### 2.2 Secondary Endpoints:

- 1. Number of acute attacks.
- 2. Time to confinement in a wheelchair.
- 3. Time to legal blindness (visual acuity of 20/200 or less in the better eye with the best correction possible).
- 4. Disability scores (disease improvement defined by at least a 1 point increase in the EDSS on consecutive evaluations at least 3 months apart).

IRB #: STU00004831-CR0001 Approved by NU IRB for use on or after 7/18/2016 through 7/17/2017.

- 5. Quality of life- SF –36.
- 6. NMO IgG aquaporin 4 autoantibody titer.

# 3.0 Background of Devic's disease

Devic's disease is similar to MS in that the body's immune system attacks the myelin surrounding nerve cells. Unlike standard MS, the attacks are not believed to be mediated by the immune system's T cells but rather by antibodies called NMO-lgG. These antibodies target a protein called aquaporin 4 in the cell membranes of astrocytes which acts as a channel for the transport of water across the cell membrane. (28) Aquaporin 4 is found in the processes of the astrocytes that surround the blood-brain barrier, a system responsible for preventing substances in the blood from crossing into the brain. The blood-brain barrier is weakened in Devic's disease, but it is currently unknown how the NMO-lgG immune response leads to demyelination.

Most research into the pathology of Devic's disease has focused on the spinal cord. The damage in the spinal cord can range from inflammatory demyelination to necrotic damage of the white and grey matter. The inflammatory lesions in Devic's disease have been classified as type II lesions (complement mediated demyelinization), but they differ from MS pattern II lesions in their prominent perivascular distribution. Therefore, the pattern of inflammation is often quite distinct from that seen in MS. (28) (33)

#### 3.1 Diagnosis

The Mayo Clinic proposed a revised set of criteria for diagnosis of Devic's disease in 2006. The new guidelines for diagnosis require two absolute criteria plus at least two of three supportive criteria being: (34)

#### Absolute criteria:

- 1. Optic neuritis
- 2. Acute myelitis

#### Supportive criteria:

- 1. Brain MRI not meeting criteria for MS at disease onset
- Spinal cord MRI with contiguous T2-weighted signal abnormality extending over 3 or more vertebral segments, indicating a relatively large lesion in the spinal cord
- NMO-IgG seropositive status. The NMO-IgG test checks the existence of antibodies against the aquaporin 4 antigen.

#### 3.1.2 Variants

After the development of the NMO-IgG test, the spectrum of disorders that comprise Devic's disease was expanded. The Devic's disease spectrum is now believed to consist of:

- Standard Devic's disease, according to the diagnostic criteria described above
  - Limited forms of Devic's disease, such as single or recurrent events of longitudinally extensive myelitis, and bilateral simultaneous or recurrent optic neuritis
  - Asian optic-spinal MS
  - Longitudinally extensive myelitis or optic neuritis associated with systemic auto-immune disease
  - Optic neuritis or myelitis associated with lesions in specific brain areas

such as the hypothalamus, periventricular nucleus, and brainstem (35)

Whether Devic's disease is a distinct disease or part of the wide spectrum of multiple sclerosis is debated. Devic's disease differs in that it usually has more severe sequelae after an acute episode than in MS, MS infrequently presents as transverse myelitis, while oligoclonal bands in the CSF, as well as white matter lesions on brain MRI, are uncommon in Devic's disease but occur in over 90% of MS patients. (36)

# 3.1.3 Proposed diagnostic criteria for neuromyelitis optica\* (76)

#### Absolute criteria:

- 1. Optic neuritis
- 2. Acute myelitis
- 3. No evidence of clinical disease outside of the optic nerve or spinal cord

#### Supportive criteria:

# Major

- 1. Negative brain MRI at onset
- 2. Spinal cord MRI with signal abnormality extending over 3 vertebral segments
- 3. CSF pleocytosis of >50 WBC/mm or > 5 neutrophils/mm

#### Minor

- 1. Bilateral optic neuritis
- 2. Severe optic neuritis with fixed visual acuity worse than 20/200 in at least one eye
- 3. Severe, fixed, attack-related weakness (MRC <2) in one or more limbs

WBC = white blood cell count; MRC = Medical Research Council

#### 3.2 Treatment of attacks

Attacks are treated with short courses of high dosage intravenous corticosteroids such as methylprednisolone IV. When attacks progress or do not respond to corticosteroid treatment, plasmapheresis can be an effective treatment. (35) Clinical trials for these treatments contain very small numbers, and most are uncontrolled.

#### 3.3 Secondary prevention

No controlled trials have established the effectiveness of treatments for the prevention of attacks. Many clinicians agree that long term immunosuppression is required to reduce the frequency and severity of attacks, while others argue the exact opposite (38). Commonly used immunosuppressant treatments include azathioprine (Imuran) plus prednisone, mycophenolate mofetil plus prednisone, Rituximab, Mitoxantrone, intravenous immunoglobulin (IVIG), and Cyclophosphamide (39) (35). The monoclonal antibody rituximab is under study (40). In 2007, Devic's disease was reported to be responsive to glatiramer acetate (41) and to low-dose corticosteroids. (42)

<sup>\*</sup>Diagnosis requires all absolute criteria and one major supportive criterion or two minor supportive criteria.

#### **Prognosis** 3.4

Normally, there is some measure of improvement in a few weeks, but residual signs and disability may persist, sometimes severely.

The disease can be monophasic, i.e. a single episode with permanent remission. However, at least 85% of patients have a relapsing form of the disease with repeated attacks of transverse myelitis and/or optic neuritis. In patients with the monophasic form the transverse myelitis and optic neuritis occur simultaneously or within days of each other. On the other hand, patients with the relapsing form are more likely to have weeks or months between the initial attacks and to have better motor recovery after the initial transverse myelitis event. Relapses usually occur early with about 55% of patients having a relapse in the first year and 90% in the first 5 years. (28) Unlike MS, Devic's disease rarely has a secondary progressive phase in which patients have increasing neurologic decline between attacks without remission. Instead, disabilities arise from the acute attacks. (28)

Approximately 20% of patients with monophasic Devic's disease have permanent visual loss and 30% have permanent paralysis in one or more legs. Among patients with relapsing Devic's disease, 50% have paralysis or blindness within 5 years. In some patients (33% in one study), transverse myelitis in the cervical spinal cord resulted in respiratory failure and subsequent death.

It is clinically important to identify risk factors that predict a relapsing course as early as possible, ideally after the NMO diagnostic criteria are met, in order that immunomodulatory therapy can be started prior to accumulation of severe neurologic deficit. It is established that female sex, older age at onset, presence of systemic autoimmunity were each independently associated with a relapsing course. Prediction of disease course is highly desirable because those with monophasic disease will not require therapeutic interventions aimed at relapse prevention. (78)

# Figure 1 Relapsing Devic's- Probability of survival



Relapsing neuromyelitis optica (NMO) survival: time from disease onset to death. Nonparametric survival curve for relapsing NMO survival. Median survival = 17.4 years. Bold line is probability estimate; lighter lines are 95 % Cl's. (76) Version Date: 07-16-2015

Devic's Disease Auto 2008


# 3.6 Epidemiology

The prevalence and incidence of Devic's disease has not been established partly because the disease is under recognized and often confused with MS (28). Devic's disease is more common in women than men, with women comprising over 2/3 of patients and more than 80% of those with the relapsing form of the disease. (28) Devic's disease is more common in Asiatic people than Caucasians. In fact, Asian optic-spinal MS (which constitutes 30% of the cases of MS in Japan) has been suggested to be identical to Devic's disease (Differences between optic-spinal and classic MS in Japanese patients). In the indigenous populations of tropical and subtropical regions, MS is rare, but when it appears it often takes the form of optic-spinal MS (43). The majority of Devic's disease patients have no affected relatives, and it is generally regarded as a non-familial condition. (28)

# 4.0 Rationale for the Proposed Treatment and Scientific Justification

The rationale for autologous HSCT of autoimmune diseases is to regenerate a new, i.e. antigen naïve immune system, from the patient's own hematopoietic stem cell. Intense immune ablation without myeloablative side effects could be accomplished with agents such as cyclophosphamide, fludarabine, and antibodies to T cells (anti-thymocyte globulin) and / or B cells (rituximab) or both T and B cells (Campath). Non-myeloablative autologous HSCT regimens are safer and pose less risk to the patient than myeloablative regimens. The initial standard non-myeloablative regimen consisted of cyclophosphamide and rabbit antithymocyte globulin (r ATG) and was pretty well tolerated. A second generation non-myeloablative regimen included cyclophosphamide and a broader and longer acting agent, Alemtuzumab, instead of r ATG. After transplantation in patients, receiving regimens, containing Alemtuzumab, potential life-threatening secondary autoimmune cytopenias, including idio pathic thrombocytopenic purpura, autoimmune neutropenia, and autoimmune hemolytic anemia, occurred late (2 to 18 months). (76)

And to date, the third generation non-myeloablative regimen, termed "Rituximab sandwich", has been well tolerated. This regimen entails 1 dose of Rituximab given before and after cyclophosphamide and r ATG.

Autologous HSCT for autoimmune diseases may be performed with either myeloablative or nonmyeloablative regimens. (74). Myeloablative regimens use cancer-specific treatments that destroy the entire marrow compartment, including marrow stem cells, resulting in irreversible and lethal marrow failure if HSCs are not reinfused. Nonmyeloablative regimens are designed specifically for autoimmune diseases, i.e., for lymphoablation without irreversible destruction of marrow stem cells. Following a nonmyeloablative regimen, hematopoietic recovery will occur without infusion of HSCs; however, autologous HSCs provide support and shorten the duration of chemotherapy-induced marrow suppression. (75).

Non-myeloablative regimen has a mortality of < 1% (table 1)

Table 1. Treatment –Related Mortality Following Autologous Hematopoietic Stem Cell Transplantation for Autoimmune Diseases (77), non-myeloablative regimen

| Source | Disease | Multicent<br>er<br>Or Single<br>Center | Treatment -Related<br>Deaths/Patients<br>No. (%) | Response |
|---|---|---|---|---|
| Burt et al | Relapsing-<br>Remitting MS | Single | 0/21 (0) | 0%progression at 2years, 62% improved |
| Craig et al | Crohn's disease | Single | 0/21 (0) | 100% remission 33% relapse |
| Oyama et al | Systemic sclerosis | Single | 0/10 (0) | 70% progression-free Survival at 2 years |
| Statkute et al | Vasculitis | Single | 0/4 (0) | Complete remission (n=3);partial response (n=1) |
| Voltarelli et<br>al | Type 1 diabetes mellitus | Single | 0/15 (0) | 13/15 patients Insulin –free |
| Vonk et al | Systemic<br>Sclerosis | Multiple | 1/26 (4) | 64% event-free Survival at 5 years |
| Burt et al | SLE | Single | 1/50 (2) | 50% disease-free Survival at 5 years |
| Snowden et al | Rheumatoid<br>Arthritis | Multiple | 0/73 (0) | 50% ACR criteria 50 or<br>Greater response in 12 m |
| Total | | | 2/200 (<1) | |

# 4.1 Selection of High Dose Immunosuppressive Therapy and Autologous HSCT Strategy for this trial

To justify any new therapy such as HSCT, the risk of dying from the disease must be higher than that expected from its treatment, or the morbidities associated with the disease must justify the treatment risks. Cyclophosphamide with or without ATG has been used to treat several patients with systemic lupus erythematosus and approximately 80 rheumatoid arthritis patients in Australia, Europe and America, again without mortality, and has been used for longer than a decade as the conditioning regimen of choice for the non-malignant disease, aplastic anemia.

At our center we have experience with a "third" generation non-myeloablative regimen termed "Rituximab sandwich" which entails 1 dose of Rituximab given before and after Cyclophosphamide and rATG, and has been used safely without unexpected toxicity.

#### Rituximab

It is chimeric murine/human monoclonal antibody to the CD20 molecule on B-lymphocytes. The molecule is combined with Fc fragment of human IgG I kappa immunoglobulin containing murine light- and heavy-chain variable region sequence and human constant region sequences. Adverse reactions caused by Rituximab include infusion reactions, mucocutaneous reactions, hypersensitivity reactions, cardiac arrhytmias and renal failure. The infusion reactions can be treated with slowing or interruption of the infusion and supportive care (diphenhydramine, acetaminophen, IV saline or vasopressors). Other reactions include: nausea, vomiting, diarrhea, headache, myalgias, arthralgias, cough, rhinitis, bronchospasm, dyspnea, sinusitis, lymphopenia, neutropenia, thrombocytopenia, anemia, abdominal pain, back pain, throat irritation, asthenia, infection. Reactivation of hepatitis B virus and progression to fulminant hepatitis has been reported in patients with negative hepatitis B surface antigen, but positive hepatitis B surface antibody.

#### Cyclophosphamide

It is a common conditioning regimen with two decades of experience in the treatment of aplastic anemia, and has been used safely without reported mortality in the treatment of autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis. Cyclophosphamide is a potent immunosuppressive agent that not only has less acute toxicity, it has less chronic side effects. Cyclophosphamide is not associated with late malignancies or cataracts

It is an alkylating agent that requires hepatic metabolism to the active metabolites, phosphoramide mustard and acrolein. These active metabolites react with nucleophilic groups. It is available as an oral or intravenous preparation. Bioavailability is 90% when given orally. The half-life of the parent compound is 5.3 hours in adults and the half-life of the major metabolite phosphoramide mustard is 8.5 hours. Liver or renal dysfunction will lead to prolonged serum half-life. CY is administered intravenously at a dosage of 60 mg/kg on each of two successive days (use adjusted ideal body weight if patient's actual body weight is greater than 100% ideal body weight). The major dose limiting side effect at high doses is cardiac necrosis. Hemorrhagic cystitis can occur and is mediated by the acrolein metabolite. This can be prevented by co-administration of MESNA or bladder

Version Date: 07-16-2015


irrigation. Other notable side effects include nausea, vomiting, alopecia, myelosuppression and SIADH. Refer to institutional manuals for more information about administration, toxicity and complications.

# Rabbit- Derived Anti-Thymocyte Globulin (r ATG)

Rabbit-derived anti-human thymocyte globulin (ATG) is a gamma globulin preparation obtained from hyperimmune serum of rabbits immunized with human thymocytes. ATG has been used predominately in solid organ transplant immunosuppressive regimens. ATG is a predominantly lymphocyte-specific immunosuppressive agent. It contains antibodies specific to the antigens commonly found on the surface of T cells. After binding to these surface molecules, ATG promotes the depletion of T cells from the circulation through mechanisms which include opsonization and complement-assisted, antibody-dependent, cell-mediated cytotoxicity. The plasma half-life ranges from 1.5-12 days. ATG is administered intravenously at a dose of 0.5 mg/kg recipient body weight on day -5 and at a dose of 1.0 mg/kg recipient body weight on days -4 and dose 1.5 mg/kg recipient body weight on days-3, -2, -1. Unlike equine ATG, rabbit ATG does not require a pre-infusion skin test to check for hypersensitivity. Methylprednisolone 250 mg will be given before every dose of ATG. Additional medications such as diphenhydramine may be given at the discretion of the attending physician. Although rare, the major toxicity is anaphylaxis; chills, fever, pruritus or serum sickness may occur.

# Method of Harvesting Stem Cells

Based on the experience of the pilot studies, the current protocol will mobilize stem cells with granulocyte-colony stimulating factor (G-CSF) and cyclophosphamide and collect stem cells by apheresis. A subsequent bone marrow harvest will be performed only if needed to supplement the peripheral blood stem cells (PBSC). Based on experience of autoimmune flares in patients receiving G-CSF alone for mobilization, patients will be mobilized with cyclophosphamide 2.0 g/m² and G-CSF 5- 10 mcg /kg.

# 5.0 Eligibility

#### 5.1 Inclusion Criteria

- 1. Age 16-65, at the time of pretransplant evaluation.
- 2. An established diagnosis of Devic's disease (more than one acute attack).
- 3. NMO- IgG aquaporin-4 autoantibody positive.

#### 5.2 Exclusion Criteria

- 1. Paraplegia or quadriplegia and legal blindness (defined as visual acuity of 20/200 or less in the better eye with the best correction possible).
- 2. Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
- Prior history of malignancy except localized basal cell, squamous skin cancer
  or carcinoma in situ of the cervix. Other malignancies for which the patient is
  judged to be cured, such as head and neck cancer, or breast cancer will be
  considered on an individual basis.
- 4. Positive pregnancy test.
- 5. Inability or unwillingness to pursue effective means of birth control. Effective birth control is defined as 1) refraining from all acts of vaginal intercourse (ABSTINENCE); 2) consistent use of birth control pills; 3) injectable birth control methods (Depo-Provera, Norplant); 4) tubal sterilization or male partner who has undergone vasectomy; 5) placement of an IUD (intrauterine device); or 6) use, with every act of intercourse, of diaphragm with contraceptive jelly and/or condoms with contraceptive foam.
- 6. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
- 7. FEV<sub>1</sub>/FVC < 60% of predicted after bronchodilator therapy (if necessary).
- 8. DLCO < 50% of predicted.
- Resting LVEF < 50 %.</li>
- 10. Serum creatinine > 2.0 mg/dl.
- 11. Known hypersensitivity to mouse, rabbit, or E. coli derived proteins.
- 12. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams.
- 13. Bilirubin > 2.0 mg/dl.
- 14. Platelet count < 100,000/up or ANC< 1000/up
- Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible.

- 16. Active infection except asymptomatic bacteriuria.
- 17. Inability to give informed consent.
- 18. HIV positive.
- 19. Transaminases > 3x of normal limits, liver cirrhosis.

# 5.3 Study Procedures

| | Baselin | During<br>Hospitaliz | First<br>100 days<br>after | 6 months<br>after<br>treatment | Every 12<br>months<br>after |
|---|---|---|---|---|---|
| | | daily | discharge<br>from<br>hospital | | treatment<br>for 5 yrs. |
| Complete history and Physical exam | Х | X | Weekly* | Х | Х |
| Disability Evaluation 9 hole peg test, timed 25- foot walk, EDSS, NRS, PASAT,MRC | Х | | X | X | X |
| MRI – Head & Spine with gadolinium | Х | | | | X<br>May do only<br>orbit & spine |
| CBC and diff | х | x | Once<br>every<br>1-2 | X | X |
| PT and PTT | Х | | | | |
| Serum chemistry | х | х | Once<br>every<br>1-2 | X | Х |
| HIV1 and HIV2 | Х | | | | |
| Serum or Urine<br>Pregnancy<br>Test | X | | | | |
| PFT w/ DLCO & FEVI/FVC | Х | | | | |
| 2 D echo | Х | | | | |
| Chest X ray | X | | <del> </del> | | |
| EKG | X | | | | |
| Urinalysis | X | | | | |
| Quantiferon Gold | X | | | | |
| TSH, T3, T4 | X | | | | |
| Serologies<br>Hepatitis A,B,C, Herpes,<br>CMV | X | | | | |

| JC virus titer | Х | | | |
|----------------------------------------------|---|---|---|---|
| QOL Questionnaires<br>SF-36 and the FACT BMT | Х | | Х | Х |
| Dental Consult | Х | | | |
| Anti-NMO | Х | ļ | Х | Х |
| Ophthalmology evaluation | Х | | | Х |

\* Until clinically stable

# 5.4 Outcome Measurement Tools - Neuropsychological, Quality of Life (QOL), a and Other Tests

All subjects will be examined (baseline) and yearly thereafter with neuropsychological exams which shall include the Paced Auditory Serial Addition Test (PASAT) and a standardized, repeatable battery of tests consisting of the Selective Reminding Test (verbal learning), 7/24 Spatial Recall Test I (visuospatial learning), and Controlled Oral Word Association (verbal fluency and semantic retrieval). These cognitive functions, in addition to the PASAT, are most often disrupted in patients with MS. Administration of these tests and MS Functional Composite (which includes timed 25-foot walk, and 9-hole peg test in addition to the PASAT) will be performed by a trained professional and should take 40 – 50 minutes. Self-administered quality of life exams (FACT-BMT and SF-36) will also be obtained pre-transplant, 6 and 12 months post-transplant, and then yearly until 5 years post-transplant.

The SF-36 (Ware 1997 and McHorney 1994) is a generic indicator of health status derived from the 245-item Medical Outcomes Study questionnaire. The SF-36 includes multi-item scales to measure the following eight dimensions; physical functioning (PF), role limitations due to physical health problems (RP), bodily pain (BP), general health perception (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and general mental health (MH). The scoring system for each dimension uses an approach which recodes the answers of each question into a 0-to-100 score, oriented so that a higher score indicates a better health state. For example, functioning scales are scored such that a high score indicates better functioning and the pain scale is scored such that a higher score indicates decreased pain. The SF-36 is a commonly used quality of life measure and facilitates comparisons across treatments and disease groups as well as against population norms.

The FACT-BMT is a valid and reliable measure of five dimensions of quality of life in a HSCT recipients (McQuellon et al BMT 1997). It consists of the 35 question Functional Assessment of Cancer Therapy (FACT) measure and a 12 question BMT subscale. It is commonly used in BMT quality of life research. Although some of the questions are specific to HSCT recipients, the vast majority of questions in the scale apply equally to patients receiving any type of therapy for their illness. Along with providing additional comparative data between treatment groups, the FACT-BMT results will allow us to study the QOL in MS patients undergoing a HSCT versus other a HSCT populations from the literature.

#### 6.0 Treatment Plan

## 6.1 Mobilization and Peripheral Blood Stem Cell Harvest:

| Day | 0 | 1 | 2 | 3 | 4 | 5 | ANC>100/ul<br>(approximately day<br>10) |
|---|---|---|---|---|---|---|---|
| Cytoxan<br>2.0 gm/m² | Х | | | | | | |
| G-CSF<br>5- | | | | | | Х | |

| 10mcg/kg/day | | |
|--------------|---|----|
| Hydration | Χ | |
| Mesna | X | |
| Apheresis | | X* |

Cytoxan dose of 2gm/m will be infused over two hours.

G-CSF- guidelines, 5-10 mcg/kg/day will be started day +5 and continued until the absolute neutrophil counts reaches at least 1,000

Hydration- guidelines, normal saline at 150-200ml/hr should be given 2 hours before cyclophosphamide and continued until 24 hours after the cyclophosphamide dose. The rate of hydration will be aggressively adjusted. BID weights will be obtained. Amount of fluid can be modified based on patient's fluid status.

Mesna, given the dose of 2.0 gm/m, infusion to be given over 24 hours.

\*Apheresis will begin when the ANC is greater than 1000/ul and continue until greater than 2.0 x 10<sup>6</sup> CD34+ cells/kg patient weight have been cryopreserved. A maximum of four apheresis will be performed. The G-CSF will continue until apheresis is discontinued.

# 6.2 Interval between Mobilization and Conditioning

In order to avoid cumulative cardiac toxicity from cyclophosphamide and to allow culture of HSC product, three weeks must separate the administration of cyclophosphamide for mobilization and for conditioning.

## 6.3 Transplant Conditioning Regimen

| Day | -7 | -6 | -5 | -4 | -3 | -2 | -1 | 0 | +1 | +6 |
|---|---|---|---|---|---|---|---|---|---|---|
| Hydration | | Х | Х | Х | X | Х | X | | | |
| Cyclophosphamide | | | Х | X | Х | X | | | | |
| 50 mg/kg/day | _ | | | | | | - | | | |
| MESNA<br>50 mg/kg/day | | | X | X | X | X | | | | |
| rATG mg/kg/day | | | 0.5 | 1.0 | 1.5 | 1.5 | 1.5 | | | |
| Stem cell reinfusion | | | | | | - 44 | | Х | | |
| Rituxan 500 mg | | X | | | | | | | X | |
| Solu-Medrol 250 mg IV | | | X | X | X | Х | X | | | |
| Apheresis catheter insertion* | X | | | | | | | | | |
| Plasmapheresis | X | | | | | | 1 | | | |

Temporary apheresis catheter placed by interventional radiology, will be removed after plasmapheresis

<u>Hydration-guidelines</u>: NS at 150-200 ml/hr should be given 2 hours before cyclophosphamide and continued until 24 hours after the last cyclophosphamide dose.

Devic's Disease Auto 2008


The rate of hydration will be aggressively adjusted. BID weights will be obtained. Amount of fluid can be modified based on patient's fluid status.

Cyclophosphamide: 50 mg/kg/day will be given IV over 2 hours in 500 cc of normal saline. If actual weight is < ideal weight, cyclophosphamide will be given based on actual weight. If actual weight is > ideal weight, cyclophosphamide will be given as adjusted weight. Adjusted weight = ideal weight + 25% (actual weight minus ideal weight).

Mesna: 50mg/day x 2 days will be given IV over 24 hours

<u>rATG</u> 0.5 mg/kg given on day –5, then 1.0 mg/kg given on day –4, then 1.5 mg/kg given on days –3 through –1. r ATG is infused over 10 hours. Premedicate with Acetaminophen 650 mg po and Diphenhydramine 25 mg po/IV 30 minutes before the infusion.

Rituxan (Rituximab) – The dose of 500 mg of Rituximab will be diluted in 500 ml 0.9 % NS and infused per standard Rituximab infusion guidelines, given on days –6 and on day + 1. Following the guidelines, Rituximab will be started at 50 mg/hr. If no reaction occurs, the dose will be increased by 50 mg/hr every 30 minutes to a maximum of 400 mg/hr.

G-CSF – guidelines, 5-10 mcg/kg/day will be started day + 5 and continued until the absolute neutrophil counts reaches at least 1,000/µl.

<u>Plasmapheresis</u>-In an autoimmune disease, the immune system attacks the body's own tissues. In many autoimmune diseases, the chief weapons of attack are antibodies, proteins that circulate in the bloodstream until they meet and bind with the target tissue. Once bound, they impair the functions of the target, and signal other immune components to respond as well.

Plasmapheresis is used to remove antibodies from the bloodstream, thereby preventing them from attacking their targets. It does not directly affect the immune system's ability to make more antibodies, and therefore may only offer temporary benefit. Neurologic diseases comprise 90% of the diseases that could profit from plasmapheresis.

Patients with clotting disorders may not be suitable candidates for plasmapheresis.

The basic procedure consists of removal of blood, separation of blood cells from plasma, and return of these blood cells to the body's circulation, diluted with fresh plasma or a substitute. Because of concerns over viral infection and allergic reaction, fresh plasma is not routinely used. Instead, the most common substitute is saline solution with sterilized human albumin protein. During the course of a single session, two to three liters of plasma is removed and replaced.

Plasmapheresis requires insertion of a venous catheter, either in a limb or central vein. Central veins allow higher flow rates and are more convenient for repeat procedures, but are more often the site of complications, especially bacterial infection.

When blood is outside the body, it must be treated to prevent it from clotting. While most of the anticlotting agent is removed from the blood during treatment, some is returned to the patient. To reduce this tendency citrate binds to calcium in the blood, calcium being essential for blood to clot. Citrate is very effective in preventing blood from clotting; however, its use can lead to life threatening low calcium levels. To prevent this complication, calcium is infused intravenously while the patient is undergoing the plasmapheresis; in addition, calcium supplementation by mouth may also be given.

Three procedures are available:

- "Discontinuous flow centrifugation." Only one venous catheter line is required.
   Approximately 300 ml of blood is removed at a time and centrifuged to separate plasma from blood cells.
- "Continuous flow centrifugation." Two venous lines are used. This method requires slightly less blood volume to be out of the body at any one time.
- "Plasma filtration." Two venous lines are used. The plasma is filtered using standard hemodialysis equipment. It requires less than 100 ml of blood to be outside the body at one time.

A single plasmapheresis session may be effective, although it is more common to have several sessions per week over the course of two weeks or more. In this case, plasmapheresis is performed at once before transplant to remove antibodies that will cause flare upon engraftment.

#### Aftercare

The patient may experience dizziness, nausea, numbness, tingling, or lightheadedness during or after the procedure. These effects usually pass quickly, allowing the patient to return to normal activities the same day.

#### Risks

Reinfusion (replacement) with human plasma may cause anaphylaxis, a life threatening allergic reaction. All procedures may cause a mild allergic reaction, leading to fever, chills, and rash. Bacterial infection is a risk, especially when a central venous catheter is used. Reaction to the citrate anticoagulant used may cause cramps and numbness, though these usually resolve on their own. Patients with impaired kidney function may require drug treatment for the effects of citrate metabolism.

Plasma contains clotting agents, chemicals that allow the blood to coagulate into a solid clot. Plasma exchange removes these. Bleeding complications are rare following plasmapheresis, but may require replacement of clotting factors (79).

# 6.4 Concurrent Treatment and Supportive Care Guidelines

#### 6.4.1 Transfusion Support Guidelines

All blood products are to be irradiated (25 Gy). CMV negative patients are to receive CMV negative blood products or alternatively (leukocyte-poor) leukofiltered blood products. Prior to administration of blood products, patients may be medicated with Benadryl 10 - 25 mg IV or po and acetaminophen 650 mg po to prevent febrile reactions.

 $\underline{\text{Red cells}}$ : For Hgb < 8.0 g/dl (Hct >27) transfuse 2 units irradiated ABO/Rh matched units.

<u>Platelets</u>: Platelets (irradiated) are given electively for platelet count less than 20  $\times$  10 $^{9}$ /l. For procedures associated with a high risk of hemorrhage, including major surgical procedures, deep tissue biopsies, lumbar puncture, placement of central vascular catheter and endoscopy of the gastrointestinal tract, maintain platelet counts greater than 50  $\times$  10 $^{9}$ /l. Platelets should be infused just before an invasive procedure. In addition to the platelet count, bleeding time, PT/PTT, fibrinogen and

other measures of coagulation may be helpful in some patients for defining the extent of any clotting dysfunction.

# 6.4.2 Infection Prophylaxis and Treatment Guidelines

All prophylactic antibiotics may be changed or discontinued according to clinical circumstances (e.g., patient allergy) as determined by the attending physician(s).

Antibacterial Prophylaxis: When neutropenia (neutrophils < 0.5 x 10<sup>9</sup>/L) occurs, prior to the development of first fever, prophylactic antibiotics will be started. Cefepime 2 grams every 8 hours or Zosyn 3.75 g IV every 4 hours is recommended. Administration of antibiotics will be done according to the institutional standard of practice of the participating center.

Antifungal Prophylaxis: Fluconazole 400 mg po daily from day of transplant until 6 months post-transplant.

Antiviral Prophylaxis: Valacyclovir or acyclovir will be administered for HSV and VZV prevention from day of transplant until 12 months post-transplant. Administration of antiviral agents will be according to the institutional standard of practice of the participating center. If there is no documented standard of practice, then administration of antibiotics will be done.

Pneumocystis carinii pneumonia (PCP) Prophylaxis: Trimethoprim-sulfamethoxazole (TMP-SMX, Bactrim) DS tablet po every Monday, Wednesday and Friday starting after engraftment (absolute neutrophil count >500/ul for 3 days) and continued for 12 months. If the patient experiences a side effect to Bactrim (e.g., rash), aerosolized pentamidine 300 mg inhaled q month for 12 months will be substituted.

#### 7.0 HOSPITAL DISCHARGE GUIDELINES

- 1. Afebrile.
- 2. No parenteral feeding required.
- 3. Platelet transfusion requirement less than 3x/week.
- 4. Neutrophil count greater than 500/ul.
- 5. Patient or family member is able to provide care.
- 6. Arrangements for follow-up with BMT physician and primary physician.

#### 8.0 SIDE EFFECTS

Risk of hematopoietic stem cell transplantation. The major hazard of this protocol is transplant-related morbidity and mortality. The marrow ablative regimen of cyclophosphamide will destroy the patient's immune/hematopoietic system and leave the patient susceptible to a wide variety of infections and bleeding complications until the reinfused stem cells engraft. Aggressive supportive care as described above will be used to prevent all avoidable risk. However, a small percentage of patients may die as a direct result of transplant related complications. Transplant related mortality is directly related to a patient's age, general medical condition, and prior exposure to prolonged or aggressive chemotherapy regimens. Transplant related complications include infections,

bleeding, venom-occlusive disease of the liver, and failure to engraft. This protocol is designed to minimize these complications.

<u>Risk of central line</u>. Placement of an external central line catheter device is a routine procedure which may be done under local or general anesthesia. Potential complications include bleeding, pneumothorax, hemothorax, or arrhythmia. Like all artificial devices, lines may become infected and require treatment with antibiotics and/or removal.

Risk of lymphopheresis and leukapheresis. This procedure requires 4-6 hours (1-2 hours for lymphopheresis) and will be performed through apheresis catheter or a 16 gauge catheter introduced into the antecubital vein. The total volume outside the body at any time does not exceed 450 ml. The most common complication is hypocalcemia arising from citrate anticoagulation, which is usually mild or rarely severe with nausea, vomiting or arrhythmias. Symptoms are avoided with replacement solutions added during apheresis, slowing the flow rate, and/or supplemental oral antacids containing calcium. Other complications are infrequent, but include hypotension, vasovagal syncope, and infection.

**Drug/chemotherapy side effects**. See Section 9 - Drug Information.

#### 9.0 DRUG INFORMATION

## 9.1 Cyclophosphamide

- 1. Other names: Cytoxan, Neosar
- 2. Chemical: 2-bis (2-chloroethyl) amino tetrahydro-2H-1, 3, 2- oxazaphosphorine-2-oxide monohydrate.
- 3. Classification: Alkylating agent.
- 4. Action: Causes prevention of cell division by forming adducts with DNA.
- 5. Metabolism: Metabolized to active compounds by microsomal enzymes in the liver. Excreted by the kidney in both the original form and as metabolites.
- 6. Availability: 25 mg and 50 mg tablets (tablets cannot be split); 100 mg, 200 mg, 500 mg, 2000 mg vials Mead Johnson and Adria.
- 7. Storage: Stable at room temperature indefinitely before reconstitution. After reconstitution, stable for 6 days upon refrigeration or for 24 hours at room temperature.
- 8. Administration: Dissolved in 500 cc 0.9%NS and administered over 60 minutes IV. Must be aggressively hydrated before, during, and for 24 hours after cyclophosphamide. If the rate of required hydration is not tolerated in a patient, bladder irrigation may need to be substituted.
- 9. Side effects: Myelosuppression, leukopenia (nadir 8-14 days), hemorrhagic cystitis, syndrome of inappropriate secretion of antidiuretic hormone (SIADH), bladder carcinoma, cellular dysplasias, mucositis, rash, alopecia, anorexia, nausea, vomiting, sterile phlebitis, rare pulmonary toxicity, teratogenicity, hemorrhage, myocarditis, infertility, secondary leukemia; with rapid IV push, oropharyngeal tingling, metallic taste, headache, urticaria, facial swelling. Metabolic abnormalities following cyclophosphamide induced cell lysis can require dialysis in patients with underlying renal insufficiency.

#### 9.2 G-CSF

- 1. Other name: Neupogen.
- 2. Description: Hematopoietic growth factor.
- 3. Drug administration: Subcutaneous administration 5-15mcg/kg/day.
- 4. Storage and Stability: 300 mcg and 480 mcg vials stored in refrigerator.
- 5. Toxicity: Myalgias, headache, flu-like symptoms, fever, bone pain in approximately 20% of patients, possible elevation of uric acid, transaminases, and LDH.

#### 9.3 ATG Rabbit

- 1. Other names: thymoglobulin
- Description: A rabbit polyclonal antibody to lymphocytes.
- Drug administration 2.0 mg/kg in D5W or NS infused over 10 hours.
- 4. Storage and Stability- 50mg/ml (5 ml ampule) vial stored in refrigerator.
- Toxicity- Side effects of ATG are serum sickness and/or anaphylaxis: chills. arthralgias, headache, myalgia, nausea, vomiting, diarrhea, chest-pain, hypotension, dyspnea, pulmonary edema, abdominal pain. Other side effects in include ab normal liver function test (SGOT, SGPT) and renal function and thrombocytopenia.

#### 9.4 Rituximab

- Other names: Rituxan
- Description : Biologic response modifier
- Action: chimeric murine/human monoclonal antibody to the CD20 molecule on Blymphocytes, the molecule is combined with Fc fragment of human IgG 1 kappa immunoglobulin containing murine light-and heavy-chain variable region sequence and human constant region sequences. Exact mechanism of action is unknown.
- 4. Availability: 10 mg/ml (10 ml and 50 ml ampules)
- Storage: protected from light at 2-8 degrees centigrade.
- 6. Administration: patients should be premedicated with 25 mg Diphenhydramine and 650 mg of Acetaminophen 30 minutes prior to each Rituximab infusion. The dose of 500 mg of Rituximab will be diluted in 500 ml of 0.9 % NS and infused per standard Rituximab infusion guidelines (start at 50 mg/hour. If no reaction occurs, increase by 50 mg/hour every 30 minutes to a maximum of 400 mg/hour).
- 7. Side effects: the most serious adverse reactions include infusion reactions, mucocutaneous reactions, hypersensitivity reactions, cardiac arrhythmias and angina. and renal failure. The infusion reactions can be treated by slowing or stopping the infusion and supportive care (Diphenhydramine, Acetaminophen, IV saline or vasopressors). Other reactions include: nausea/vomiting/diarrhea, headache. bronchospasm, dyspnea, myalgias. arthralgias, cough, rhinitis. lymphopenia, leucopenia, neutropenia, thrombocytopenia, anemia, abdominal pain, back pain, throat irritation, asthenia, infection. Reactivation of hepatitis B virus and progression to fulminant hepatitis has been reported in patients with negative hepatitis B surface antigen, but positive hepatitis B surface antibody.

#### **Evaluation of toxicity** 10.0

Daily assessment will be made with regards to toxicity by one of the protocol investigators. Common Toxicity Criteria Scale will be used to grade all non-hematologic toxicities. Version Date: 07-16-2015

# 11.0 Adverse event reporting

Any serious <u>unexpected</u> event <u>or</u> any death during the study, regardless of the cause, must be immediately reported to Richard K. Burt (312-695-4960). The Toxicity Grading for adverse events is according to NCI common toxicity criteria for adverse events (CTCAE) version 2.0 at website http://ctep.info,nih.gov

# 11.1 To be reported by phone (312-695-4960) or FAX (312-695-4961) to Richard Burt:

a) All lethal (Grade 5) reactions. This information is to be immediately reported to Dr. Burt who will report it within 72 hours of a working day to the IRB and FDA.

# 11.2 To be reported in writing within 10 working days:

- a) Grade 3 or 4 reactions, except myelosuppression which is anticipated. These will be reported by Dr. Burt on annual reports to the FDA
- b) Any death within 30 days of study treatment, even if patient is off study.

# 12.0 Evaluation of response

To be performed at 6 months post-transplant, and then every year for 5 years.

# 13.0 Number of patients - 40, for phase I /II study.

# 14.0 Data Management

Collection of data, management, data checking and verification, will be performed by the PI and his team at Northwestern University Medical School. General Clinical Research Center statistician Dr. Jovanovic will be available to assist with data management and analysis. Analysis will be performed by the research staff using S-Plus, SAS and Microsoft Excel.

#### 15.0 Statistical references

Cox DR: Regression models and life tables (with discussion). Journal of the Royal Statistical Society, B, 74, 187-220. 1972.

Kaplan EL, Meier P: Nonparametric estimation from incomplete observations. Journal of the American Statistical Association, 53, 457-81. 1958.

## 16.0 Criteria for removal from study

- 1. Pregnancy prior to starting therapy.
- 2. Patient withdrawal before beginning conditioning regimen or after successful recovery of hematopoiesis.
- 3. Disease progression making travel and follow-up studies of such inconvenience that they impose a significant risk or burden to the patient.

Devic's Disease Auto 2008


# 17.0 Follow- up procedures for withdrawal subjects

Unless the patient refuses, subjects who withdraw from the study will be followed in a manner consistent with the monitoring plan.

# 18.0 Stopping rules

Study will be held for any treatment –related death until reviewed and approved by the IRB, DSMB, and the US FDA. A treatment related death is any death deemed possibly, probably, or definitely related to therapy.

Disease relapse or progression will not be defined as toxicity but disease progression or relapse in greater than 5 of 10 patients having return of active Devic's within 1 year of treatment will also trigger stopping of the study until reviewed by IRB, FDA, and DSMB. Triggering of stopping rules will prompt cessation of new enrollment, notification of the IRB and FDA and performance of a comprehensive safety review.

# 19.0 Records to be kept

Records will be kept in the office of the Division of Immunotherapy.

#### 20.0 References

- Civin CI, Almeida-Porada G, Lee MJ, Olweus J, Terstappen LW, Zanjani ED. Sustained, retransplantable, multilineage engraftment of highly purified adult human bone marrow stem cells in vivo. *Blood* 1996, 88(11): 4102-9.
- 2. De Koning J, Van Bekkum DW, Dicke KA, Dooren LJ, Radl J, Van Rood JJ. Transplantation of bone-marrow cells and fetal thymus in an infant with lymphopenic immunological deficiency. *Lancet* 1969, 1(7608): 1223-7.
- Ikehara S, Yasumizu R, Inaba M, Izui S, Hayakawa K, Sekita K, Toki J, Sugiura K, Iwai H, Nakamura T. Long-term observations of autoimmune-prone mice treated for autoimmune disease by allogeneic bone marrow transplantation. *Proceedings of the National Academy of Sciences of the United States of America* 1989, 86(9): 3306-10.
- Ikehara S, Ohtsuki H, Good RA, Asamoto H, Nakamura T, Sekita K, Muso E, Tochino Y, Ida T, Kuzuya H. Prevention of type I diabetes in nonobese diabetic mice by allogenic bone marrow transplantation. *Proceedings of the National Academy of Sciences of the United States of America* 1985, 82(22): 7743-7.
- LaFace DM, Peck AB. Reciprocal allogeneic bone marrow transplantation between NOD mice and diabetes-nonsusceptible mice associated with transfer and prevention of autoimmune diabetes. *Diabetes* 1989, 38(7): 894-901.
- 6. Kamiya M, Sohen S, Yamane T, Tanaka S. Effective treatment of mice with type II collagen induced arthritis with lethal irradiation and bone marrow transplantation. *Journal of Rheumatology* 1993, 20(2): 225-30.
- Pestronk A, Drachman DB, Teoh R, Adams RN. Combined short-term immunotherapy for experimental autoimmune myasthenia gravis. *Annals of Neurology* 1983, 14(2): 235-41.
- 8. VanBekkum DW. Conditioning regimens for the treatment of experimental arthritis with autologous bone marrow transplantation. *Bone Marrow Transplantation* 2000, 25(4): 357-64.
- 9. van Bekkum DW, Bohre EP, Houben PF, Knaan-Shanzer S. Regression of adjuvant-induced arthritis in rats following bone marrow transplantation. *Proceedings of the National Academy of Sciences of the United States of America* 1989, 86(24): 10090-4.
- 10. Karussis DM, Vourka-Karussis U, Lehmann D, Ovadia H, Mizrachi-Koll R, Ben-Nun A, Abramsky O, Slavin S. Prevention and reversal of adoptively transferred, chronic relapsing experimental autoimmune encephalomyelitis with a single high dose cytoreductive treatment followed by syngeneic bone marrow transplantation. *Journal of Clinical Investigation* 1993, 92(2): 765-72.
- van Gelder M, Kinwel-Bohre EP, van Bekkum DW. Treatment of experimental allergic encephalomyelitis in rats with total body irradiation and syngeneic BMT. Bone Marrow Transplantation 1993, 11(3): 233-41.

- 12. Burt RK, Burns W, Ruvolo P, Fischer A, Shiao C, Guimaraes A, Barrett J, Hess A. Syngeneic bone marrow transplantation eliminates V beta 8.2 T lymphocytes from the spinal cord of Lewis rats with experimental allergic encephalomyelitis. *Journal of Neuroscience Research* 1995, 41(4): 526-31.
- Nakamura T, Good RA, Yasumizu R, Inoue S, Oo MM, Hamashima Y, Ikehara S. Successful liver allografts in mice by combination with allogeneic bone marrow transplantation. Proceedings of the National Academy of Sciences of the United States of America 1986, 83(12): 4529-32.
- 14. Gandy KL, Weissman IL. Tolerance of allogeneic heart grafts in mice simultaneously reconstituted with purified allogeneic hematopoietic stem cells. *Transplantation* 1998, 65(3): 295-304.
- 15. van Gelder M, van Bekkum DW. Effective treatment of relapsing experimental autoimmune encephalomyelitis with pseudoautologous bone marrow transplantation. *Bone Marrow Transplantation* 1996, 18(6): 1029-34.
- Burt RK, Padilla J, Begolka WS, Canto MCD, Miller SD. Effect of disease stage on clinical outcome after syngeneic bone marrow transplantation for relapsing experimental autoimmune encephalomyelitis. *Blood* 1998, 91(7): 2609-16.
- 17. Miller SD, Gerety SJ. Immunologic aspects of Theiler's murine encephalomyelitis virus (TMEV)-induced demyelinating disease. *Semin. Virol* 1990, 1: 263-272.
- Miller SD, Vanderlugt CL, Begolka WS, Pao W, Yauch RL, Neville KL, Katz-Levy Y, Carrizosa A, Kim BS. Persistent infection with Theiler's virus leads to CNS autoimmunity via epitope spreading. *Nature Medicine* 1997, 3(10): 1133-6.
- Burt RK, Padilla J, Dal Canto MC, Miller SD. Viral hyperinfection of the central nervous system and high mortality after hematopoietic stem cell transplantation for treatment of Theiler's murine encephalomyelitis virus-induced demyelinating disease. *Blood* 1999, 94(8): 2915-22.
- 20. Mancardi GL, Saccardi R, Filipppi M, et al. Autologous hempatopoietic stem cell transplantation suppresses gd-enhanced MRI activity in MS. *Neurology* 2001, 57: 62-68.
- 21. Burt RK, Traynor AE, Cohen B, Karlin KH, Davis FA, Stefoski D, Terry C, Lobeck L, Russell EJ, Goolsby C, Rosen S, Gordon LI, Keever-Taylor C, Brush M, Fishman M, Burns WH. T cell-depleted autologous hematopoietic stem cell transplantation for multiple sclerosis: Report on the first three patients. *Bone Marrow Transplantation* 1998, 21(6): 537-41.
- 22. Burt RK, Traynor AE, Pope R, Schroeder J, Cohen B, Karlin KH, Lobeck L, Goolsby C, Rowlings P, Davis FA, Stefoski D, Terry C, Keever-Taylor C, Rosen S, Vesole D, Fishman M, Brush M, Mujias S, Villa M, Burns WH. Treatment of autoimmune disease by intense immunosuppressive conditioning and autologous hematopoietic stem cell transplantation. *Blood* 1998, 92(10): 3505-14.
- 23. Openshaw H, Stuve O, Antel JP, Nash R, Lund BT, Weiner LP, Kashyap A, McSweeney P, Forman S. Multiple sclerosis flares associated with recombinant granulocyte colony-stimulating factor. *Neurology* 2000, 54(11): 2147-50.

- 24. Burt RK, Fassas A, Snowden J, van Laar JM, Kozak T, Wulffraat N, Nash R, Dunbar CE, Arnold R, Prentice G, Bingham S, Marmont A, McSweeney P. Collection of hematopoietic stem cells from patients with autoimmune diseases. *Bone Marrow Transplantation*, 2001; 28, 1-12.
- 25. Holmberg LA, Boeckh M, Hooper H, Leisenring W, Rowley S, Heimfeld S, Press O, Maloney DG, McSweeney P, Corey L, Maziarz RT, Appelbaum FR, Bensinger W. Increased incidence of cytomegalovirus disease after autologous CD34-selected peripheral blood stem cell transplantation. *Blood* 1999, 94(12): 4029-35.
- 26. Openshaw H, Lund BT, Kashyap A, Atkinson R, Sniecinski I, Weiner LP, Forman S. Peripheral blood stem cell transplantation in multiple sclerosis with busulfan and cyclophosphamide conditioning: Report of toxicity and immunological monitoring. *Biology of Blood & Marrow Transplantation* 2000, 6(5A): 563-75.
- Pittock SJ, Weinshenker BG, Lucchinetti CF, Wingerchuk DM, Corboy JR, Lennon VA (2006). "Neuromyelitis optica brain lesions localized at sites of high aquaporin 4 expression". Arch. Neurol. 63 (7): 964–8. doi:10.1001/archneur.63.7.964. PMID 16831965.
- 28. Wingerchuk, DM (2006). "Neuromyelitis optica". The International MS Journal 13: 42-50. PMID 16635421.
- 29. Lennon VA, Wingerchuk DM, Kryzer TJ, et al (2004). "A serum autoantibody marker of neuromyelitis optica: distinction from multiple sclerosis". Lancet 364 (9451): 2106–12. doi:10.1016/S0140-6736(04)17551-X. PMID 15589308.
- Pittock SJ, Lennon VA, Krecke K, Wingerchuk DM, Lucchinetti CF, Weinshenker BG (2006). "Brain abnormalities in neuromyelitis optica". *Arch. Neurol.* 63 (3): 390–6. doi:10.1001/archneur.63.3.390. PMID 16533966.
- 31. Lennon VA, Kryzer TJ, Pittock SJ, Verkman AS, Hinson SR (2005). "IgG marker of optic-spinal multiple sclerosis binds to the aquaporin-4 water channel". J. Exp. Med. 202 (4): 473–7. doi:10.1084/jem.20050304. PMID 16087714.
- 32. Mayo Clinic. Devic's Disease Symptoms. Retrieved on 2008-03-11.
- 33. Lucchinetti CF, Mandler RN, McGavern D, et al (2002). "A role for humoral mechanisms in the pathogenesis of Devic's neuromyelitis optica". *Brain* 125 (Pt 7): 1450–61. PMID 12076996.
- 34. Wingerchuk DM, Lennon VA, Pittock SJ, Lucchinetti CF, Weinshenker BG (2006). "Revised diagnostic criteria for neuromyelitis optica". *Neurology* 66 (10): 1485–9. doi:10.1212/01.wnl.0000216139.44259.74. PMID 16717206.
- 35. Wingerchuk, Dean (2006). "Neuromyelitis Optica (Devic's Syndrome)". 2006 Rare Neuroimmunologic Disorders Symposium. Retrieved on 2007-01-05.
- 36. Pearce JM (2005). "Neuromyelitis optica". *Spinal Cord* 43 (11): 631–4. Devic's Disease Auto 2008 29 of 56 Version Date: 07-16-2015

- doi:10.1038/sj.sc.3101758. PMID 15968305.
- 37. Cree BA, Goodin DS, Hauser SL (2002). "Neuromyelitis optica". Seminars in neurology 22 (2): 105–22. doi:10.1055/s-2002-36534. PMID 12524556.
- 38. Poser CM, Brinar VV (2007). "Disseminated encephalomyelitis and multiple sclerosis: two different diseases a critical review". *Acta Neurol. Scand.* 116 (4): 201–6. doi:10.1111/j.1600-0404.2007.00902.x. PMID 17824894.
- 39. Weinstock-Guttman B, Ramanathan M, Lincoff N, et al (2006). "Study of mitoxantrone for the treatment of recurrent neuromyelitis optica (Devic disease)". Arch. Neurol. 63 (7): 957–63. doi:10.1001/archneur.63.7.957. PMID 16831964.
- Matiello M, Jacob A, Wingerchuk DM, Weinshenker BG (2007). "Neuromyelitis optica". *Curr. Opin. Neurol.* 20 (3): 255-60. doi:10.1097/WCO.0b013e32814f1c6b. PMID 17495617.
- Gartzen K, Limmroth V, Putzki N (2007). "Relapsing neuromyelitis optica responsive to glatiramer acetate treatment". Eur. J. Neurol. 14 (6): e12-3. doi:10.1111/j.1468-1331.2007.01807.x. PMID 17539924.
- 42. Watanabe S, Misu T, Miyazawa I, et al (2007). "Low-dose corticosteroids reduce relapses in neuromyelitis optica: a retrospective analysis". doi:10.1177/1352458507077189. PMID 17623727.
- 43. Cabre P, Signate A, Olindo S, et al (2005). "Role of return migration in the emergence of multiple sclerosis in the French West Indies". *Brain* 128 (Pt 12): 2899–910. doi:10.1093/brain/awh624. PMID 16183661.
- 44. T. Jock Murray (2005). *Multiple Sclerosis: The History of a Disease*. New York: Demos Medical Publishing. ISBN 1888799803.
- 45. Devic's Disease Research Mayo Clinic. Retrieved on 2007-11-22.
- 46. Lennon, V., Kryzer T., Pittock S., Verkman A., Hinson S. (2005), "IgG marker of optic-spinal multiple sclerosis binds to the aquaporin-4 water channel". JEM, Volume 2002, number 4,473-477
- 47. Wingerchuk, DM (2006). "Neuromyelitis optica". The International MS Journal 13: 42-. PMID 16635421.
- 48. Samijn JP, te Boekhorst PA, Mondria T; et al. Intense T cell depletion followed by autologous bone marrow transplantation for severe multiple sclerosis. *J Neurol Neurosurg Psychiatry*. 2006; 77(1):46-50.
- 49. Oyama Y, Barr WG, Statkute L; et al. Autologous non-myeloablative hematopoietic stem cell transplantation in patients with systemic sclerosis. *Bone Marrow Transplant*. 2007; 40(6):549-555.
- 50. Statkute L, Oyama Y, Barr WG; et al. Autologous non-myeloablative hematopoietic stem

- cell transplantation for refractory systemic vasculitis [published online ahead of print October 18, 2007]. *Ann Rheum Dis.* doi:10.1136/ard.2007.070227. ABSTRACT
- 51. Voltarelli JC, Couri CE, Stracieri AB; et al. Autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. *JAMA*. 2007; 297(14):1568-1576.
- 52. Vonk MC, Marjanovic Z, van den Hoogen FH; et al. Long-term follow-up results after autologous haematopoietic stem cell transplantation for severe systemic sclerosis [published online ahead of print May 25, 2007]. *Ann Rheum Dis.* doi:10.1136/ard.2007.071464. 2008; 67(1):98-104.
- 53. Burt RK, Traynor A, Statkute L; et al. Nonmyeloablative hematopoietic stem cell transplantation for systemic lupus erythematosus. *JAMA*. 2006; 295(5):527-535.
- 54. Oyama Y, Craig RM, Traynor AE; et al. Autologous hematopoietic stem cell transplantation in patients with refractory Crohn's disease. *Gastroenterology*. 2005; 128(3):552-563.
- 55. Snowden JA, Passweg J, Moore JJ; et al. Autologous hematopoietic stem cell transplantation in severe rheumatoid arthritis: a report from the EBMT and ABMTR. *J Rheumatol.* 2004; 31(3):482-488.
- Al-toma A, Visser OJ, van Roessel HM; et al. Autologous hematopoietic stem cell transplantation in refractory celiac disease with aberrant T cells. *Blood.* 2007; 109(5):2243-2249.
- 57. Ouyang J, Zhu WH, Wang C, Chen B. Autologous hematopoietic stem cell transplantation for progressive multiple sclerosis: report of efficacy and safety at three yr of follow up in 21 patients. *Clin Transplant.* 2006; 20(4):485-489.
- 58. Xu J, Ji BX, Su L, Dong HQ, Sun XJ, Liu CY. Clinical outcomes after autologous haematopoietic stem cell transplantation in patients with progressive multiple sclerosis. *Chin Med J (Engl)*. 2006; 119(22):1851-1855.
- 59. Capello E, Saccardi R, Murialdo A; et al, Italian GITMO-Neuro Intergroup on ASCT for Multiple Sclerosis. Intense immunosuppression followed by autologous stem cell transplantation in severe multiple sclerosis. *Neurol Sci.* 2005; 26(suppl 4):S200-S203.
- 60. Carreras E, Saiz A, Marín P; et al. CD34+ selected autologous peripheral blood stem cell transplantation for multiple sclerosis: report of toxicity and treatment results at one year of follow-up in 15 patients. *Haematologica*. 2003; 88(3):306-314.
- 61. Fassas A, Passweg JR, Anagnostopoulos A; et al, Autoimmune Disease Working Party of the EBMT (European Group for Blood and Marrow Transplantation). Hematopoietic stem cell transplantation for multiple sclerosis: a retrospective multicenter study. *J Neurol*. 2002; 249(8):1088-1097. [Published correction appears in *J Neurol*. 2002; 249(11)1619].

- 62. Kozák T, Havrdová E, Pit'ha J; et al. High-dose immunosuppressive therapy with PBPC support in the treatment of poor risk multiple sclerosis. *Bone Marrow Transplant*. 2000; 25(5):525-531.
- 63. Burt RK, Cohen BA, Russell E; et al. Hematopoietic stem cell transplantation for progressive multiple sclerosis: failure of a total body irradiation-based conditioning regimen to prevent disease progression in patients with high disability scores. *Blood*. 2003; 102(7):2373-2378.
- 64. Nash RA, Bowen JD, McSweeney PA; et al. High-dose immunosuppressive therapy and autologous peripheral blood stem cell transplantation for severe multiple sclerosis. *Blood*. 2003; 102(7):2364-2372.
- 65. Openshaw H, Lund BT, Kashyap A; et al. Peripheral blood stem cell transplantation in multiple sclerosis with busulfan and cyclophosphamide conditioning: report of toxicity and immunological monitoring. *Biol Blood Marrow Transplant*. 2000; 6(5A):563-575.
- 66. Daikeler T, Kötter I, Bocelli Tyndall C; et al, EBMT Autoimmune Diseases Working Party. Haematopoietic stem cell transplantation for vasculitis including Behcet's disease and polychondritis: a retrospective analysis of patients recorded in the European Bone Marrow Transplantation and European League Against Rheumatism databases and a review of the literature. Ann Rheum Dis. 2007; 66(2):202-207.
- 67. Saccardi R, Kozak T, Bocelli-Tyndall C; et al, Autoimmune Diseases Working Party of EBMT. Autologous stem cell transplantation for progressive multiple sclerosis: update of the European Group for Blood and Marrow Transplantation autoimmune diseases working party database. *Mult Scler.* 2006; 12(6):814-823.
- 68. De Kleer IM, Brinkman DM, Ferster A; et al. Autologous stem cell transplantation for refractory juvenile idiopathic arthritis: analysis of clinical effects, mortality, and transplant related morbidity. *Ann Rheum Dis.* 2004; 63(10):1318-1326.
- 69. Farge D, Passweg J, van Laar JM; et al. Autologous stem cell transplantation in the treatment of systemic sclerosis: report from the EBMT/EULAR registry. *Ann Rheum Dis.* 2004; 63(8):974-981.
- 70. Jayne D, Passweg J, Marmont A; et al, European Group for Blood and Marrow Transplantation, European League Against Rheumatism Registry. Autologous stem cell transplantation for systemic lupus erythematosus. *Lupus*. 2004; 13(3):168-176.
- 71. Binks M, Passweg JR, Furst D; et al. Phase I/II trial of autologous stem cell transplantation in systemic sclerosis: procedure related mortality and impact on skin disease. *Ann Rheum Dis.* 2001; 60(6):577-584.
- 72. Montoto S, Canals C, Rohatiner AZ; et al, EBMT Lymphoma Working Party. Long-term follow-up of high-dose treatment with autologous haematopoietic progenitor cell support in 693 patients with follicular lymphoma: an EBMT registry study [published online ahead of print July 19, 2007]. Leukemia. doi:10.1038/sj.leu.2404850. 2007; 21(11):2324-2331.
- 73. Brown JR, Feng Y, Gribben JG; et al. Long-term survival after autologous bone marrow transplantation for follicular lymphoma in first remission. *Biol Blood Marrow Transplant*. Devic's Disease Auto 2008 32 of 56 Version Date: 07-16-2015

- 2007; 13(9):1057-1065.
- 74. Nash RA, McSweeney PA, Crofford LJ; et al. High-dose immunosuppressive therapy and autologous hematopoietic cell transplantation for severe systemic sclerosis: long-term follow-up of the US multicenter pilot study. *Blood*. 2007; 110(4):1388-1396.
- 75. Burt RK, Marmont A, Oyama Y; et al. Randomized controlled trials of autologous hematopoietic stem cell transplantation for autoimmune diseases: the evolution from myeloablative to lymphoablative transplant regimens. *Arthritis Rheum.* 2006; 54(12):3750-3760.
- 76. Statkute L, Verda L, Oyama Y; et al. Mobilization, harvesting and selection of peripheral blood stem cells in patients with autoimmune diseases undergoing autologous hematopoietic stem cell transplantation. *Bone Marrow Transplant*. 2007; 39(6):317-329.
- 77. Wingerchuk: Neurology, Volume 60(5).March 11, 2003.848-853
- Richard K. Burt; Yvonne Loh; William Pearce; Nirat Beohar; Walter G. Barr; Robert Craig;
   Yanting Wen; Jonathan A. Rapp; John Kessler Clinical Applications of Blood-Derived and
   Marrow-Derived Stem Cells for Nonmalignant Diseases. *JAMA*. 2008; 299(8):925–936.
- 79. Wingerchuk DM, Weinshenker BG. Neurology, 2003 Mar 11;60 (5):848-53. Neuromyelitis optica: clinical predictors of a relapsing course and survival.
- 80. Samuels, Martin, and Steven Feske, editors. Office Practice of Neurology. New York: Churchill Livingstone, 1996.

## Appendix I

Muscle strength testing scale MRC - Scale

- 0: total lack of voluntary contraction
- 1: trace faint contraction without any movement
- 2: poor contraction with very weak movement through full range of movement, when gravity is eliminated.
- 3: fair contraction with movement through the complete joint, range against gravity.
- 4: good contraction with full range of movement against gravity and some resistance.
- 5: normal contraction with normal strength through full range of motion against full resistance.

# Appendix II

#### **KURTZKE EDSS - Extended Disability Status Scale (EDSS) (41)**

- 0= Normal neurological exam (all grade 0 in Function Systems (FS); Cerebral grade 1 acceptable).
- 1.0= No disability, minimal signs in one FS (i.e., grade 1 excluding Cerebral grade1).
- 1.5= No disability minimal signs in more than one S (more than one grade 1 excluding Cerebral grade 1).
- 2.0= Minimal disability in one FS (one FS grade 2, other 0 or 1).
- 2.5= Minimal disability in two FS (two FS grade 2, other 0 or 1).
- 3.0= Moderate disability in one FS (one FS grade 3, other 0 or 1), or mild disability in three or four FS (three/four FS grade 2, other 0 or 1) though fully ambulatory.
- 3.5= Fully ambulatory but with moderate disability in one FS (one grade 3) and one or two FS grade 2; or two FS grade 3; or Five FS grade 2 (others 0 or 1).
- 4.0= Fully ambulatory without aid, self-sufficient, up and about some 12 hours a day despite relatively severe disability consisting of one FS grade 4 (others 0 or 1), or combinations of lesser grades exceeding limits of previous steps. Able to walk without aid or rest some 500 meters.
- 4.5= Fully ambulatory without aid, up and about much of the day, able to work a full day, may otherwise have some limitation of full activity or require minimal assistance; characterized by relatively severe disability, usually consisting of one FS grade 4 (others 0 or 1) or combinations of lesser grades exceeding limits of previous steps. Able to walk without aid or rest for some 300 meters.
- 5.0= Ambulatory without aid or rest for about 200 meters; disability sever enough to impair full daily activities (e.g. to work full day without special provisions). (Usual FS equivalents are one grade 5 alone, others 0 or 1; or combinations of lesser grades usually exceeding specifications for step 4.0)
- 5.5= Ambulatory without aid or rest for about 100 meters; disability severe enough to preclude full daily activities. (Usual FS equivalents are one grade 5 alone, others 0 or 1; or combinations of lesser grades usually exceeding those for step 4.0).
- 6.0= Intermittent or unilateral constant assistance (cane, crutch or brace) required to walk about 100 meters with or without resting. (Usual FS equivalents are combinations with more than two FS grade 3+).
- 6.5= Constant bilateral assistance (cane, crutch, or brace) required to walk about 20 meters without resting. (Usual FS equivalents are combinations with more than two FS grade 3+).
- 7.0= Unable to walk beyond about 5 meters even with aid, essentially restricted to wheelchair, wheels self in standard wheelchair and transfers alone; up and about in w/c some 12 hours a day. (Usual FS equivalents are combinations with more than one FS grade 4+; very rarely, pyramidal grade 5 alone).
- 7.5= Unable to take more than a few steps; restricted to wheelchair, may need aid in transfer, wheels self but cannot carryon in standard wheelchair a full day; may require motorized wheelchair. (Usual FS equivalents are combinations with more than one FS grade 4+).
- 8.0= Essentially restricted to bed or chair or perambulated in wheelchair, but may be out of bed itself much of the day; retains many self-care functions; generally has effective use of arms. (Usual FS equivalents are combinations, generally grade 4+ in several systems).
- 8.5= Essentially restricted to bed much of the day; has some effective use of arm (s); retains some self-care functions. (Usual FS equivalents are combinations, generally 4+ in several systems).
- 9.0= Helpless bed patient; can communicate and eat. (Usual FS equivalents are combinations, mostly grade 4+).
- 9.5= Totally helpless bed patient; unable to communicate effectively or eat/swallow. (Usual FS equivalents are combinations, almost all grade 4+).
- 10.0= Death due to MS

#### **FUNCTIONAL SYSTEMS**

#### Pyramidal functions

- 0= Normal
- 1= Abnormal signs without disability
- 2= Minimal disability
- 3= Mild or moderate paraparesis or hemiparesis; severe monoparesis
- 4= Marked paraparesis or hemiparesis; moderate quadriparesis; or monoplegia
- 5= Paraplegia, hemiplegia, or marked quadriparesis
- 6= Quadriplegia
- V= Unknown

## **Cerebellar Functions**

- 0= Normal
- 1= Abnormal signs without disability
- 2= Mild ataxia
- 3= Moderate truncal or limb ataxie
- 4= Severe ataxia; all limbs
- 5= Unable to perform coordinated movements due to ataxia
- V= Unknown
- X= Is used throughout after each number when weakness (grade 3 or more on pyramidal) interferes with testing.

#### **Brain Stem Functions**

- 0= Normal
- 1= Signs only
- 2= Moderate nystagmus or other mild disability
- 3= Severe nystagmus, marked extraocular weakness, or moderate disability of other cranial nerves
- 4= Marked dysarthria or other marked disability
- 5= Inability to swallow or speak
- V= Unknown

#### **Sensory Functions**

- 0= Normal
- 1= Vibration or figure-writing decrease only, in one or two limbs
- 2= Mild decrease in touch or pain or position sense and/or moderate decrease in vibration in one or two limbs; or vibratory (c/s figure writing) decrease alone in three or four limbs.
- 3= Moderate decrease in touch or pain or position sense, and/or essentially lost vibration in one or two limbs; or mild decrease in touch or pain and/or moderate decrease in all proprioceptive tests in three or four limbs.

- 4= Marked decrease in touch or pain or loss of proprioception, alone or combined, in one or two limbs; or moderate decrease in touch or pain and/or severe proprioceptive decrease in more than two limbs
- Loss (essentially) of sensation in one or two limbs; or moderate decrease in touch or pain and/or loss of proprioception for most of the body below the head
- 6= Sensation essentially lost below the head
- V= Unknown

#### **Bowel and Bladder Functions**

- 0= Normal
- 1= Mild urinary hesitancy, urgency, or retention
- 2= Moderate hesitancy, urgency, retention of bowel or bladder, or rare urinary incontinence
- 3= Frequent urinary incontinence
- 4= In need of almost constant catheterization
- 5= Loss of bladder function
- 6= Loss of bowel and bladder function
- V= Unknown

## Visual (or Optic) Functions

- 0= Normal
- 1= Scotoma with visual acuity (corrected) better than 20/30
- 2= Worse eye with scotoma with maximal visual acuity (corrected) or 20/30 to 20/59
- 3= Worse eye with large scotoma, or moderate decrease in fields, but with maximal visual acuity (corrected) of 20/60 to 20/99
- Worse eye with marked decrease of fields and maximal visual acuity (corrected) of 20/100 to 20/200; grade 3 plus maximal acuity of better eye of 20/60 or less
- 5= Worse eye with maximal visual acuity (corrected) less than 20/200; grade 4 plus maximal acuity of better eye of 20/60 or less

- 6= Grade 5 plus maximal visual acuity of better eye of 20/60 or less
- V= Unknown

X= Is added to grades 0 to 6 for presence of temporal pallor

# Cerebral (or Mental) Functions

- 0≡ Normal
- 1= Mood alteration only (Does not affect DSS score)
- 2= Mild decrease in mentation
- 3= Moderate decrease in mentation
- 4= Marked decrease in mentation (chronic brain syndrome moderate)
- 5= Dementia or chronic brain syndrome severe or incompetent
- V= Unknown

#### **Other Functions**

- 0= None
- 1= Any other neurologic findings attributed to MS (specify)
- V= Unknown

# **EDSS WORKSHEET**

| | <br>1 | |
|---------------|-------|-------------------|
| Date | | |
| Pyramidal | | |
| Cerebellar | | |
| Brainstem | | is and the second |
| Sensory | | |
| Bowel/Bladder | | |
| Visual | | |
| Mental | | |
| Other | | |
| EDSS | | |

Appendix III
SCRIPPS NEUROLOGICAL RATING SCALE (NRS) WORKSHEET\*

| | MAXIMUM | | DEGREE OF IMPAIRMENT | | |
|---|---|---|---|---|---|
| SYSTEMS EXAMINED | POINTS | NORMAL | MILD | MOD. | SEVERE |
| Mentation and Mood | 10 | 10 | 7 | 4 | 0 |
| Cranial Nerves: | 21 | | | | |
| Visual Acuity | | 5 | 3 | 1 | 0 |
| Fields, Discs, Pupils | | 6 | 4 | 2 | 0 |
| Eye Movements | | 5 | 3 | 1 | 0 |
| Nystagmus* | | 5 | 3 | 1 | 0 |
| Lower Cranial Nerves | 5 | 5 | 3 | 1 | 0 |
| Motor: | 20 | | | | |
| RU | | 5 | 3 | 1 | 0 |
| LU | | 5 | 3 | 1 | 0 |
| RL | | 5 | 3 | 1 | 0 |
| LL | | 5 | 3 | 1 | 0 |
| DTRS: | 8 | | | | |
| UE | | 4 | 3 | 1 | 0 |
| LE | | 4 | 3 | 1 | 0 |
| Babinski: R:L (2 ea) | 4 | 4 | - | • | 0 |
| Sensory: | 12 | | | | |
| RU | ļ | 3 | 2 | 1 | 0 |
| LU | | 3 | 2<br>2<br>2 | 1 | 0 |
| RL | | 3 | | 1 | 0 |
| LL | | 3 | 2 | 1 | 0 |
| Cerebellar: | 10 | | | | |
| UE | | 5 | 3 | 1 | 0 |
| LE | | 5 | 3 | 1 | 0 |
| Gait: Trunk & Balance | 10 | 10 | 7 | 4 | 0 |
| Special Category: | 0 | 0 | -3 | -7 | -10 |
| Bladder/Bowel/Sexual | ľ | | | | |
| Dysfunction | | | | | |
| TOTALS | 100 | | | | |

<sup>\*</sup>Points assigned for each component of the neurologic examination are subtotaled and points for autonomic dysfunction are subtracted leaving the final (NRS) score.

| <b>NEUROLOGICAL RATING SCALE SCORE:</b> |
|-----------------------------------------|

# **Appendix IV**

**PASAT** 





Lotal Connect trans



Devic's Disease Auto 2008


FORMS FOR THE MULTIPLE SCLEROSIS PUNCTIONAL COMPOSITE

#### COUNTRY FUNCTIONS PASAT FORMER Nibox ID Narlet PASAT - Form B 2 - 2N 6 KALLEL 1 10 13 4) 13 165 111 13 SCC ) ij. 11 2, 3 ġ, 4 43 1 \$3 ΙÚ 13 Ž. 71 G. S 4 1 ς 12 Ó 12 $\tfrac{5}{2}-\tfrac{1}{4}$ 5 3 -<u>i</u> 4 N 43 13 1 1 1.4 .7 ij Ĝ ţ J. Ė $C_{\delta}^{k}$ Ś si i i . di 1. Ď N Ð 111 Į6 Lotal Correct (raw) 7-8 7 RAH: #2 3 6 15 1-1 43 (i)1.4 10 1 (Court 5 ă, 63 S Éì 1.0 11 1 4 2 8 š 3 $\cdot \bar{\delta}$ 10 \* } : \$ h 7 13 Š, Ġ S

Version Date: 07-16-2015

11)

11

| | 1684 | S FOR THE MILITIPLE | SCLEROSIS FUNCTIONAL COMPOSI |
|---|---|---|---|
| - COCHTAL DINCTON | PASATS | (INISTARY SCORE | 511 I |
| Subject 170 Number Solve | - The second sec | { \$ 2.5 } | V - 1 2 2 2 |
| PASA | E<br>f Summ | ary Score She | ef |
| FORM USED (Check one) | | Lund & President | Purm B |
| PASAT 3" | Value | Range | |
| Total Correct for a completed PASA4-3% econology cocum | states that | n-60<br>Historian patient | Pertermane. |
| | A44. | B/4 | |
| It PASA'T 3" was not completed four Cong | ¥1 | Specify | |
| (ii) Unable to complete trial due to physical in | allitationes | | |
| Ch. Chber 14 | | | |
| PASAT 2" | Value | Range | |
| letal Correct | | 0.40 | |
| or as completed PASA L27, sectors any currents | tages that 3 | flected the patient sq | ferfansa mig |
| (PASAL 2" was not completed (mark an)) | | Specifi | |
| (1) I habile to complete trial due to physical la | | Spens | |
| T. They • | naanens 🤏 | BM Fish. | |
| a 5,431% 2 | | | |
| id it take more than one attempt to get one succe<br>ses, please specify reason or for more than one i<br>getentiates some space and | satist tradit. E<br>trempte d seja | 3 Yes C1 No<br>d) | |
| PANAT3" | PAS | 112" | |
| brial correct in first built | | correct in Sea half<br>correct in second half | |
| Hal Commission Corrects | | esting sering entire en- | 10 |
| oral emission errors | 7.4.1 | office of critical | |



Appendix V

SF-36




| Name | | _ |
|---------------------|------------|---------------|
| Date of Transplant_ | | <del></del> - |
| | Visit Date | |

# Short Form- 36 Health Survey (SF-36)

**INSTRUCTIONS:** The survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities.

Answer every question by marking the answer as indicated. If you are unsure about how to answer a question, please give the best answer you can.

| 1. | In general, would you say your health is: (circle one) | |
|---|---|---|
| a. | Excellent | 1 |
| b. | Very Good | 2 |
| c. | Good | 3 |
| d. | Fair | 4 |
| e. | Poor | 5 |
| 2. | COMPARED TO ONE YEAR AGO, how would you rate y | our health in general NOW? |
| | The state of the state of the would you rate y | our health in general NOW: |
| | Much better now than one year ago | - |
| a. | | 1 |
| a.<br>b. | Much better now than one year ago | 2 |
| a.<br>b.<br>c. | Much better now than one year ago Somewhat better now than one year ago | 2 |



# 3. The following items are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

Circle one number on each item

| | ACTIVITIES | Yes,<br>Limited<br>A Lot | Yes,<br>Limited<br>A Little | No<br>Not<br>Limited<br>At All |
|---|---|---|---|---|
| a. | Vigorous activities, such as running, lifting | 1 | 2 | 3 |
| b. | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf. | 11 | 2 | 3 |
| c. | Lifting or carrying groceries. | 11 | 2 | 3 |
| d. | Climbing several flights of stairs. | 1 | 2 | 3 |
| e. | Climbing one flight of stairs. | 1 | 2 | 3 |
| f. | Bending, kneeling, or stooping. | 1 | 2 | 3 |
| g. | Walking more than a mile. | 1 | 2 | 3 |
| h. | Walking several blocks. | 1 | 2 | 3 |
| i. | Walking one block. | 1 | 2 | 3 |
| i. | Bathing or dressing yourself. | 1 | 2 | 3 |



| 4. | During the past 4 weeks, have you had any of the follow<br>regular daily activities as a result of your physical heal | ving proble<br>th? | ems with yo | our work or of |
|---|---|---|---|---|
| | Circle one number on each line | | | |
| a. | Cut down on the amount of time you spent on work or other activities. | | YES 1 | NO<br>2 |
| b. | Accomplished less than you would like. | ••••• | 1 | 2 |
| c. | Were limited in the kind of work or other activities. | | 1 | 2 |
| d. | Had difficulty performing the work or other activities (for example, it took extra effort). | | 1 | 2 |
| 5. | During the past 4 weeks, have you had any of the follow<br>work or other regular daily activities as a result of any e<br>(such as feeling depressed or anxious)? | ing proble<br>emotional p | ms with you<br>problems | ur |
| | work or other regular daily activities as a result of any o | ing proble | ms with you<br>problems | ur |
| | work or other regular daily activities as a result of any e (such as feeling depressed or anxious)? | ing proble<br>emotional p<br>YES | ms with you<br>problems<br>NO | ur |
| Cir | work or other regular daily activities as a result of any e (such as feeling depressed or anxious)? | emotional p | oroblems<br>NO | ur |
| Cir<br>a. | work or other regular daily activities as a result of any of (such as feeling depressed or anxious)? The cole one number on each line. Cut down on the amount of time you spent on work or | emotional p YES | NO 2 | ur |

| 6. | probl | ng the past 4 weeks, to what extent has your physical health or emo<br>ems interfered with your normal social activities with family, frien<br>bors, or groups? | tional<br>ds, |
|---|---|---|---|
| | Circle | one | |
| | a. | Not at all | 1 |
| | b. | Slightly | 2 |
| | c. | Moderately | 3 |
| | d. | Quite a bit | 4 |
| | e. | Extremely | 5 |
| 7. | How r | nuch bodily pain have you had during the past 4 weeks? | |
| | a. | None | 1 |
| | | Very mild | 2 |
| | c. | Mild | 3 |
| | | Moderate | 4 |
| | e. | Severe | 5 |
| | f. | Very Severe | 6 |

| 8. | | g the past 4 weeks, how much did pain ding both work outside the home and h | | | u <b>r n</b> orn | nal wor | ·k | |
|---|---|---|---|---|---|---|---|---|
| | ` | | , | | Circle o | ne | | |
| | a. | Not at all | | | | | 1 | |
| | b. | Slightly | | | | | 2 | |
| | | Moderately | | | | | 3 | |
| | | Quite a bit | | | | | 4 | |
| | | Extremely | | | | | 5 | |
| 9. | during | questions are about how you feel and he the past 4 weeks. For each question, p closest to the way you have been feeling | lease give | | | • | | |
| | How m | nuch of the time during the past 4weeks | | | A | | A | |
| | (circle o | one) | All of<br>the<br>Time | Most of the Time | Good<br>Bit of<br>Time | Some<br>of the<br>Time | Little<br>of the<br>Time | None<br>of the<br>Time |
| a. | Did yo | ou feel full of pep? | 1 | 2 | 3 | 4 | 5 | 6 |
| b. | Have y | ou been a very nervous person? | 1 | 2 | 3 | 4 | 5 | 6 |
| c. | | ou felt so down in the dumps thatg could cheer you up? | 1 | 2 | 3 | 4 | 5 | 6 |
| d. | Have y | ou felt calm and peaceful? | 1, | 2 | 3 | 4 | 5 | 6 |
| e. | Did yo | u have a lot of energy? | 1 | 2 | 3 | 4 | 5 | 6 |
| f. | Have y | ou felt downhearted and blue? | 1 | 2 | 3 | 4 | 5 | 6 |
| g. | Did yo | u feel worn out? | 1 | 2 | 3 | 4 | 5 | 6 |
| h. | Have y | ou been a happy person? | 1 | 2 | 3 | 4 | 5 | 6 |
| i | Did vo | u feel tired? | 1 | 2 | 2 | 4 | _ | _ |

| emoti | ng the past 4 weeks, how much of the tin<br>onal problems interfered with your socie<br>ves, etc.)? | | | | |
|---|---|---|---|---|---|
| Telati | , | | | Circle | one |
| a. | All of the time | | | | .1 |
| b. | Most of the time | | | | 2 |
| c. | Some of the time | | *************************************** | | .3 |
| d. | A little of the time | | ****** | | .4 |
| e. | None of the time | | | | .5 |
| | TRUE or FALSE is <i>each</i> of the followin<br>number on each line) Definitely True | | or you?<br>Don't<br>Know | Mostly<br>False | Definitely<br>False |
| | I seem to get sick a little easier 1 than other people. | | | | |
| c. | I am healthy as anybody I know. 1 | 2 | 3 | 4 | 5 |
| d. | I expect my health to get worse. 1 | 2 | 3 | 4 | 5 |
| e. | My health is excellent. 1 | 2 | 3 | 4 | 5 |
| I confirm that | the information on this survey is accurate | Patient's initials: | Date: | | |



# **Appendix VI**

#### **FACT BMT**





# FACT - BMT (VERSION 3)

Below is a list of statements that other people with your illness have said are important. By circling one number per line, please indicate how true each statement has been for you during the past 7 days.

#### **PHYSICALWELL-BEING**

| Dur | ing the past 7 days: | Not at<br>All | A Little<br>Bit | Some-<br>what | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|---|
| 1. | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| 2. | I have nausea | 0 | 1 | 2 | 3 | 4 |
| 3. | Because of my physical condition, I have | | | | | |
| | trouble meeting the needs of my family | 0 | 1 | 2 | 3 | 4 |
| 4. | I have pain | 0 | 1 | 2 | 3 | 4 |
| 5. | I am bothered by side effects of treatment | 0 | 1 | 2 | 3 | 4 |
| 6. | I feel sick | 0 | 1 | 2 | 3 | 4 |
| 7. | I am forced to spend time in bed | 0 | 1 | 2 | 3 | 4 |

8. Looking at the above 7 questions, how much would you say your

PHYSICAL WELL-BEING affects your quality of life?

(Circle one number)

0 1 3 5 Not at all

10 Very much so

#### **SOCIAL/FAMILYWELL-BEING**

| During the past 7 days: Very at All Bit what a Bit Much | Not | A Little | Some- | Quite | |
|---|---|---|---|---|---|
| 9. I feel distant from my friends | 0 | 1 | 2 | 3 | 4 |
| 10. I get emotional support from my family | 0 | 1 | 2 | 3 | 4 |
| 11. I get support from my friends and neighbors | 0 | 1 | 2 | 3 | 4 |
| 12. My family has accepted my illness | 0 | 1 | 2 | 3 | 4 |
| 13. Family communication about my illness is poor | 0 | 1 | 2 | 3 | 4 |
| 14. I feel close to my partner (or the person who | | | | | |
| is my main support) | 0 | 1 | 2 | 3 | 4 |
| 15. Have you been sexually active during the | | | | | |
| past year? D No D Yes | | | | | |
| If "Yes": I am satisfied with my sex life | 0 | 1 | 2 | 3 | 4 |
| 16. Looking at the above 7 questions, how much would ye | ou say yo | ur | | | |

**SOCIAL/FAMILY WELL-BEING** affects your quality of life?

(Circle one number)

Not at all

10 Very much so



Study SC00-02-FactBMTg (2/02) Page 1 of 3

# RELATIONSHIP WITH DOCTOR

| During the past 7 days: | Not<br>at Ali | A Little<br>Bit | Some-<br>what | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|
| 17. I have confidence in my doctor(s) | 0 | 1 | 2 | 3 | 4 |
| 18. My doctor is available to answer my questions | 0 | 1 | 2 | 3 | 4 |
| 19. Looking at the above 2 questions, how much would | | | | | |
| RELATIONSHIP WITH THE DOCTOR affects your qu | uality of life | ? (Circle | one numb | er) | |
| 0 1 2 3 4 5 6 7 8 9 | 9 10 | | | | |
| Not at all Ve | ery much so | | | | |

# **EMOTIONALWELL-BEING**

| Duri | ing the past 7 days: | Not at | A Little<br>Bit | Some-<br>what | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|---|
| 20. | I feel sad | 0 | 1 | 2 | 3 | 4 |
| 21. | I am proud of how I'm coping with my illness | 0 | 1 | 2 | 3 | 4 |
| 22. | I am losing hope in the fight against my illness | 0 | 1 | 2 | 3 | 4 |
| 23. | I feel nervous | 0 | 1 | 2 | 3 | 4 |
| 24. | I worry about dying | 0 | 1 | 2 | 3 | 4 |
| 25. | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| 26. | Looking at the above 6 questions, how much would you | say yo | ur | | | |
| EMO | TIONALWELL-BEING affects your quality of life? | | (Circ | le one nur | nber) | |
| | 0 1 2 3 4 5 6 7 8 9<br>Not at all Very | 10<br>much so | ) | | | |

#### **FUNCTIONALWELL-BEING**

| Dur | ing the past 7 days: | Not at<br>All | A Little<br>Bit | Some-<br>what | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|---|
| 27. | I am able to work (include work in home) | 0 | 1 | 2 | 3 | 4 |
| 28. | My work (include work in home) is fulfilling | 0 | 1 | 2 | 3 | 4 |
| 29. | I am able to enjoy life | 0 | i | 2 | 3 | 4 |
| 30. | I have accepted my illness | 0 | 1 | 2 | 3 | 4 |
| 31. | I am sleeping well | 0 | 1 | 2 | 3 | 4 |
| 32. | I am enjoying the things I usually do for fun | 0 | 1 | 2 | 3 | 4 |
| 33. | I am content with the quality of my life right now | 0 | 1 | 2 | 3 | 4 |
| 34. | Looking at the above 7 questions, how much would you | ı say yo | ur | | | |
| TUN | CTIONAL WELL-BEING affects your quality of life? | | (Circ | le one nu | nber) | |
| | 0 1 2 3 4 5 6 7 8 9 | 10 | | | - | |
| | Not at all Very | much so | ) | | | |

Devic's Disease Auto 2008


# **ADDITIONAL CONCERNS**

| Dur | ing the past 7 days: | Not at<br>All | A Little<br>Bit | Some-<br>what | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|---|
| 35. | I am concerned about keeping my job | | | | | |
| | (Include work in home) | 0 | 1 | 2 | 3 | 4 |
| 36. | I feel distant from other people | 0 | 1 | 2 | 3 | 4 |
| 37. | I worry that the transplant will not work | 0 | 1 | 2 | 3 | 4 |
| 38. | The effects of treatment are worse than | | | | | |
| | I had imagined | 0 | 1 | 2 | 3 | 4 |
| 39. | I have a good appetite | 0 | 1 | 2 | 3 | 4 |
| 40. | I like the appearance of my body | 0 | 1 | 2 | 3 | 4 |
| 41. | I am able to get around by myself | 0 | 1 | 2 | 3 | 4 |
| 42. | I get tired easily | 0 | 1 | 2 | 3 | 4 |
| 43. | I am interested in having sex | 0 | 1 | 2 | 3 | 4 |
| 44. | I have concerns about my ability to have children | 0 | 1 | 2 | 3 | 4 |
| 45. | I have confidence in my nurse(s) | 0 | 1 | 2 | 3 | 4 |
| 46. | I regret having the bone marrow transplant | 0 | 1 | 2 | 3 | 4 |
| 47. | Looking at the above 12 questions, how much would yo | u say y | our | | | |
| ADD: | ITIONAL CONCERNS affects your quality of life? | . • | (Circ | le one nun | nber) | |
| | 0 1 2 3 4 5 6 7 8 9 10 | | | | | |

Not at all Very much so